CLINICAL TRIAL: NCT06754891
Title: A Phase Ib Clinical Trial to Evaluate the Efficacy and Safety of TQH3906 in Adults With Moderately to Severely Active Ulcerative Colitis or Crohn's Disease
Brief Title: Clinical Trial of TQH3906 Capsules for the Treatment of Adult Patients With Moderately to Severely Active Ulcerative Colitis or Crohn's Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQH3906-Ib-01
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQH3906 capsules (Experimental): Administration of TQH3906 capsules for 8 weeks
  Interventions: Drug: TQH3906 capsules

INTERVENTIONS:
Drug: TQH3906 capsules — TQH3906 is an allosteric inhibitor targeting kinase.

SUMMARY:
This is an open-label, single-arm Phase Ib exploratory study, divided into Cohort 1: moderate to severe active ulcerative colitis, and Cohort 2: moderate to severe active Crohn's disease. Each cohort is divided into two phases. The first phase mainly explores the safety and tolerability of three dose groups of TQH3906 (12mg, 24mg, and 32mg). Based on the findings of the first phase, the second phase of the study will be conducted to select 1-2 dose groups for preliminary efficacy confirmation in ulcerative colitis and Crohn's disease. The subjects will take TQH3906 capsules orally for 8 weeks to evaluate the safety, efficacy, and pharmacokinetic (PK) characteristics of TQH3906 capsules in subjects with moderate to severe active ulcerative colitis or Crohn's disease. The study will include a screening period of up to 4 weeks, an 8-week treatment period, and a 4-week follow-up period after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years (inclusive of both 18 and 75), regardless of gender.
* Diagnosed with ulcerative colitis or Crohn's disease for ≥3 months, as assessed by histological or endoscopic examination prior to screening.
* Active moderate to severe UC or CD. .
* Subjects must have failed at least one of the following drug treatments for UC or CD or be intolerant: oral aminosalicylates, oral corticosteroids, immunosuppressants, biologics, etc.
* If subjects are using the following drugs for UC or CD at the time of screening, their treatment should be stabilized with oral aminosalicylates for at least 3 weeks before the first dose of the trial medication, or stabilized with oral systemic corticosteroids for at least 2 weeks before the first dose of the trial medication, and maintain a stable dose during the trial period.
* Subjects (including partners) are willing to voluntarily take appropriate and effective contraceptive measures from the time of screening until 3 months after the last administration of the study medication.
* Before the trial, understand in detail the nature, significance, potential benefits, possible inconveniences, and potential risks of the trial, understand the research procedures, and voluntarily sign the informed consent form.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Subjects diagnosed with indeterminate colitis, radiation colitis, or ischemic colitis.
* Have severe complications such as local stenosis, intestinal obstruction, intestinal perforation, lower gastrointestinal bleeding, intestinal cancer or tendency towards cancer, toxic megacolon; rectal colon polyps and anal diseases, etc., as assessed by the investigator, may affect the subject's efficacy and safety assessment.
* Subjects currently have a stoma, ileal pouch-anal anastomosis, fistula, and according to the physician's judgment, may require surgery or drug intervention within 12 weeks of entering the study, or may require ileostomy or colostomy.
* Subjects have had a large segment of the small intestine resected (>100cm) or have been diagnosed with short bowel syndrome, or subjects require total parenteral nutrition.
* Subjects have a recorded positive test for Clostridium difficile toxin (C. difficile) in stool or positive polymerase chain reaction (PCR) test. If the result is positive, subjects may be re-screened after appropriate treatment and re-tested no earlier than 7 days after the end of treatment.
* Abnormal serum virology during the screening period: a) Active hepatitis, or positive for Hepatitis B surface antigen (HBsAg) and positive for hepatitis B virus (HBV)-DNA, or positive for Hepatitis B core antibody (HBcAb) and positive for HBV-DNA, or positive for hepatitis B virus (HCV) antibodies and positive for HCV-RNA; b) Positive for HIV antibodies during the screening period, or history of HIV infection; c) Positive for Treponema pallidum antibodies and positive for non-treponemal serologic tests (RPR or TRUST) during the screening period.
* History of active tuberculosis during the screening period or latent tuberculosis infection (defined as enzyme-linked immunospot assay (T-SPOT) positive without clinical manifestations). (Note: Patients with latent tuberculosis infection may be re-screened after starting preventive treatment for one month according to the guidelines. To continue participating in the study, patients must agree to complete the preventive treatment plan during the study period, but rifampin treatment should be avoided.)
* History of severe herpes zoster or herpes simplex infection, including but not limited to herpes encephalitis, disseminated herpes simplex, and generalized herpes zoster.
* History of severe bacterial, fungal, or viral infections within 2 months before the first dose requiring hospitalization and intravenous antibiotic or antiviral treatment.
* Received live vaccines within 4 weeks before the first dose or plan to receive live vaccines during the study period.
* Clinically significant infections during the screening period, including but not limited to upper respiratory tract infections, lower respiratory tract infections, herpes simplex, herpes zoster, requiring antibiotic or antiviral treatment.
* Subjects with any major illness or unstable clinical condition (such as kidney, liver, blood, gastrointestinal, endocrine, lung, mental, neurological, immune, or local active infection/infectious diseases), as determined by the investigator, are not suitable for participating in this study.
* Abnormal laboratory tests during the screening period: a) alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3 times the upper limit of normal (ULN); b) Hemoglobin <90g/L; c) White blood cell count <3.0×109/L; d) Neutrophil count <1.0×109/L; e) Lymphocyte count <0.5×109/L; f) Platelet count <100×109/L; g) Total bilirubin >2 times ULN; h) Other significant laboratory test abnormalities that the investigator considers the subject unsuitable for participation in this study.
* Subjects with poorly controlled diabetes or diabetes with significant complications (such as retinopathy or nephropathy).
* History of malignant tumors (including in situ carcinoma) and lymphoproliferative diseases within 5 years before the first dose.
* Received any marketed or investigational biologics within 8 weeks before the first dose or 5 half-lives (whichever is longer).
* Received small molecule drugs such as Upadacitinib, Ozanimod, or other marketed or investigational drugs within 4 weeks or 5 half-lives (whichever is longer) before the first dose.
* Received fecal microbiota transplantation, cyclosporine, tacrolimus, mycophenolate mofetil, thalidomide, or other drugs within 4 weeks before the first dose.
* Received any other investigational drugs within 1 month or 5 half-lives (whichever is longer) before the first dose.
* Underwent surgical procedures within 4 weeks before the first dose or plan to undergo surgical procedures during the study period.
* Received immunoglobulins or blood products within 4 weeks before the first dose.
* Used potent CYP450 inducers (such as rifampin, phenobarbital, carbamazepine, phenytoin sodium, etc.) within 4 weeks before the first dose.
* Used local treatments (enemas or suppositories), intravenous steroids, azathioprine or 6-mercaptopurine, anti-UC or CD Chinese medicine, anti-infective drugs, or anti-diarrheal drugs within 2 weeks before the first dose.
* Subjects receiving methotrexate treatment must not have received methotrexate treatment for the current course within at least 42 days before screening, or stable-dose methotrexate treatment within at least 28 days before the first dose.
* Received nonsteroidal anti-inflammatory drug (NSAID) treatment within 1 week before the first dose (except for topical NSAIDs and low-dose aspirin for cardiovascular protection).
* Subjects who have undergone organ transplantation and require ongoing immunosuppressive treatment.
* Allergic to any known components of TQH3906, or with any history of severe drug allergies.
* History of drug abuse or positive urine drug screening.
* Any other reasonable medical, psychiatric, or social reasons that the investigator considers the subject unable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | Baseline up to week 16
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Clinical remission rate: Ulcerative colitis (UC): Mayo score | Week 8
  UC: Mayo score ≤2 and no single item score >1.
Clinical remission rate: Ulcerative colitis (UC): Crohn's disease (CD) | Week 8
  Crohn's disease: Average daily stool frequency ≤2.8 and average daily abdominal pain score ≤1, with neither exceeding the baseline score.

SECONDARY OUTCOMES:
The change in Inflammatory Bowel Disease Questionnaire (IBDQ) score | Week 8
  The change in Inflammatory Bowel Disease Questionnaire (IBDQ) score relative to the baseline. Improvement ≥16points.
Peak concentration (Cmax) | Day 1: within 1 hour pre-dose, 1, 2, 3, 4, 6, 8, 12, and 24 hours post dose; within 1 hour pre-dose on Day 15, 29, 57, Day 57: 1, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  Maximum plasma drug concentration of study drug.
Plasma concentration at steady state (Cav, SS) | Day 1: within 1 hour pre-dose, 1, 2, 3, 4, 6, 8, 12, and 24 hours post dose; within 1 hour pre-dose on Day 15, 29, 57, Day 57: 1, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  The plasma concentration at which the rate of administration and rate of elimination are in equilibrium.
Clinical Response Rate: UC: A decrease of ≥2 points and ≥30% from the baseline in the Mayo score | Week 8
  UC: A decrease of ≥2 points and ≥30% from the baseline in the Mayo score, as well as a decrease of ≥1 point in the rectal bleeding score (RBS) from the baseline or an absolute RBS value of ≤1.
Clinical Response Rate: Crohn's disease: A reduction of at least 100 points in the Crohn's disease activity index | Week 8
  Crohn's disease: A reduction of at least 100 points in the Crohn's disease activity index from the baseline.
Endoscopic Remission: UC: The endoscopy subscore in the Mayo score | Week 8
  UC: The endoscopy subscore in the Mayo score is 0 or 1 point.
Endoscopic Remission: CD: The Simple endoscopic score for Crohn's disease (SES-CD) score | Week 8
  CD: The SES-CD score is ≤4 and has decreased by at least 2 points from the baseline, with no subscore of any individual variable being >1.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The First Affilliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - First affiliated hospital of guangzhou medical university, Guangzhou, Guangdong
  - Luoyang First People's Hospital, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hosiptal, Tongji Medical College, Huazhong University of Science And Technolocy, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital Of University Of South China, Hengyang, Hunan
  - The first hospital of Jilin University, Changchun, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan